CLINICAL TRIAL: NCT04830267
Title: A Phase II Randomized Trial of Camrelizumab With Stereotactic Body Radiotherapy Versus Camrelizumab Alone in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: The Efficacy of Camrelizumab Plus Stereotactic Body Radiotherapy in R/M NPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ying Wang, Associate Director of Chongqing University Cancer Hospital, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Camresbrt
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Camrelizumab; Stereotactic body radiotherapy; R/M NPC; Best overall response
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; spartalizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab alone (Active Comparator): Camrelizumab 200mg IV every 2 weeks
  Interventions: Drug: Camrelizumab
- Stereotactic body radiotherapy plus Camrelizumab (Experimental): Stereotactic body radiotherapy 27Gy/3F and Camrelizumab 200mg IV every 2 weeks
  Interventions: Drug: Camrelizumab; Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg IV starting day 1 and then every 2 weeks thereafter. Treatment with Camrelizumab will continue until progression or unacceptable toxicity.
  Other Names: Anti-PD-1 antibody
Radiation: Stereotactic body radiotherapy — Image guided, stereotactic body radiotherapy (27 Gy over 3 fractions given every other day) to a single lesion to start by study day 14 (study day 1 is day of first dose of Camrelizumab).
  Other Names: SBRT
  Arms: Stereotactic body radiotherapy plus Camrelizumab

SUMMARY:
Camrelizumab is an antibody targeting programmed death receptor 1 (PD-1) and its ligand programmed death-ligand 1 (PD- L1) that is designed to boost the immune system. It does this by allowing immune cells to fight the cancer. Stereotactic body radiotherapy is a potential immunostimulatory therapy that may amplify antitumor response when combined with camrelizumab.

DETAILED DESCRIPTION:
All eligible patients from 3 hospitals will be equally randomized between the 2 following treatment groups:

Standard treatment group: Camrelizumab 200mg IV every 2 weeks. Experimental group: Stereotactic body radiotherapy 27Gy/3F and Camrelizumab 200mg IV every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines.
3. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study obligations.
4. Target Population:

   Males and females ≥ 18 years of age Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2. Histologically confirmed metastatic or recurrent nasopharyngeal carcinoma.
5. Subjects must have at least two lesions:

   At least one lesion must be safely amenable to irradiation. This can be a lesion that was previously irradiated as long as prior radiation was at least 6 months prior to projected first fraction of SBRT and as long as reirradiation dose constraints are being met.

   A separate, not-to-be-irradiated lesion measurable by CT or MRI per RECIST 1.1 criteria.
6. The peripheral blood EBV DNA copy number can be obtained.
7. Prior palliative or curative radiotherapy must be completed at least 14 days prior to randomization.
8. Immunosuppressive doses of systemic medication, such as steroids or absorbed topical steroids (doses >10mg/day prednisone or equivalent) must be discontinued at least 14 days prior to Camrelizumab administration.
9. Screening laboratory values must meet the following criteria (using CTCAE v4.0) and should be obtained within 28 days prior to randomization:

   WBC ≥ 2 K/microliter Neutrophils ≥ 1.5 K/microliter Platelets ≥ 100 K/microliter Hemoglobin ≥ 9.0 g/deciliter Serum Creatinine ≤ 1.5 x ULN or creatinine clearance > 40ml/min using the Cockcroft-Gault formula.

   Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL AST/ALT ≤ 3 x ULN Total bilirubin <1.5 x ULN (except subjects with Gilbert Syndrome who can have total bilirubin <3.0 mg/deciliter).

   Subjects must have a resting baseline O2 saturation by pulse oximetry of >=92% at rest.
10. Reproductive Status:

Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 28 days prior to randomization.

Women must not be breastfeeding Women of childbearing potential must agree to follow instructions for method(s) of contraception from time of enrollment for the duration of treatment with Camrelizumab plus 5 half- lives plus 30 days for a total of 23 weeks post treatment completion.

Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving Camrelizumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product.

Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception.

Azoospermic males and women of childbearing potential who are continuously not heterosexually active are exempt from contraceptive requirements. However, they still must have a pregnancy test.

Exclusion Criteria:

1. Target Disease Exceptions:

   Active brain metastases (untreated brain metastases or growth on imaging as defined below) or leptomeningeal disease are not allowed. Subjects with brain metastases are eligible if these have been treated and there is no MRI (or CT if MRI contraindicated) evidence of progression for at least 8 weeks after treatment for these metastases is complete and within 28 days prior to first study treatment.
2. Medical History and Concurrent Diseases:

   Any medical disorder that, in the opinion of the investigator, might increase the risk associated with study participation or interferes with the interpretation of study results.

   Prior active malignancy within the previous 3 years except for locally curable cancers such as basal or squamous skin cancer, superficial bladder, low risk prostate cancer, breast, or cervix cancer. If other prior malignancy was active within prior 3 years, enrollment requires approval of a principal investigator.

   Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration should be excluded. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
3. Physical and Laboratory Test Findings:

   Positive test for hepatitis B virus surface antigen or hepatitis C virus ribonucleic acid indicating acute or chronic infection.

   Known history of testing positive for HIV or known AIDS. Any grade 4 laboratory abnormalities. Allergies and Adverse Drug Reaction History of allergy to Camrelizumab components History of severe hypersensitivity reaction to any monoclonal antibody.
4. Prohibited or Restricted Treatments:

The following medications are prohibited during the study:

Immunosuppressive agents (except to treat a drug-related adverse event). Systemic corticosteroids > 10 mg daily prednisone equivalent save for exclusion outlined in the below paragraphs.

Any concurrent chemotherapy, hormonal therapy, immunotherapy, or investigational agents for treatment of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Best overall response (BOR) | Time Frame: 96 weeks
  As determined by the investigator using RECIST 1.1 criteria between patients receiving Camrelizumab and stereotactic body radiotherapy and those receiving Camrelizumab alone. BOR rate is defined as the number of patients randomized to a given arm with a best overall response of complete response (CR) or partial response (PR) of non-irradiated lesions divided by the total number of patients randomized to the given arm. In order to ascertain this endpoint, efforts will be made so that patients will be followed for 96 weeks or until progression of disease (and treatment cessation), whichever comes first. At each time-point, subjects should have CT/MR of neck, chest, abdomen, and pelvis with contrast.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Ph.D, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (3):
- China (3):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Wanzhou, Chongqing Municipality
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDermott DF, Shah R, Gupte-Singh K, Sabater J, Luo L, Botteman M, Rao S, Regan MM, Atkins M. Quality-adjusted survival of nivolumab plus ipilimumab or nivolumab alone versus ipilimumab alone among treatment-naive patients with advanced melanoma: a quality-adjusted time without symptoms or toxicity (Q-TWiST) analysis. Qual Life Res. 2019 Jan;28(1):109-119. doi: 10.1007/s11136-018-1984-3. Epub 2018 Sep 6. PMID 30191365
- [Background] Janjigian YY, Bendell J, Calvo E, Kim JW, Ascierto PA, Sharma P, Ott PA, Peltola K, Jaeger D, Evans J, de Braud F, Chau I, Harbison CT, Dorange C, Tschaika M, Le DT. CheckMate-032 Study: Efficacy and Safety of Nivolumab and Nivolumab Plus Ipilimumab in Patients With Metastatic Esophagogastric Cancer. J Clin Oncol. 2018 Oct 1;36(28):2836-2844. doi: 10.1200/JCO.2017.76.6212. Epub 2018 Aug 15. PMID 30110194
- [Background] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452
- [Background] Burnette BC, Liang H, Lee Y, Chlewicki L, Khodarev NN, Weichselbaum RR, Fu YX, Auh SL. The efficacy of radiotherapy relies upon induction of type i interferon-dependent innate and adaptive immunity. Cancer Res. 2011 Apr 1;71(7):2488-96. doi: 10.1158/0008-5472.CAN-10-2820. Epub 2011 Feb 7. PMID 21300764
- [Background] Sharma A, Bode B, Studer G, Moch H, Okoniewski M, Knuth A, von Boehmer L, van den Broek M. Radiotherapy of human sarcoma promotes an intratumoral immune effector signature. Clin Cancer Res. 2013 Sep 1;19(17):4843-53. doi: 10.1158/1078-0432.CCR-13-0352. Epub 2013 Jul 16. PMID 23861514
- [Background] Deng L, Liang H, Burnette B, Beckett M, Darga T, Weichselbaum RR, Fu YX. Irradiation and anti-PD-L1 treatment synergistically promote antitumor immunity in mice. J Clin Invest. 2014 Feb;124(2):687-95. doi: 10.1172/JCI67313. Epub 2014 Jan 2. PMID 24382348
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Background] Golden EB, Demaria S, Schiff PB, Chachoua A, Formenti SC. An abscopal response to radiation and ipilimumab in a patient with metastatic non-small cell lung cancer. Cancer Immunol Res. 2013 Dec;1(6):365-72. doi: 10.1158/2326-6066.CIR-13-0115. PMID 24563870
- [Background] Zandberg DP, Strome SE. The role of the PD-L1:PD-1 pathway in squamous cell carcinoma of the head and neck. Oral Oncol. 2014 Jul;50(7):627-32. doi: 10.1016/j.oraloncology.2014.04.003. Epub 2014 May 10. PMID 24819861
- [Background] McBride S, Sherman E, Tsai CJ, Baxi S, Aghalar J, Eng J, Zhi WI, McFarland D, Michel LS, Young R, Lefkowitz R, Spielsinger D, Zhang Z, Flynn J, Dunn L, Ho A, Riaz N, Pfister D, Lee N. Randomized Phase II Trial of Nivolumab With Stereotactic Body Radiotherapy Versus Nivolumab Alone in Metastatic Head and Neck Squamous Cell Carcinoma. J Clin Oncol. 2021 Jan 1;39(1):30-37. doi: 10.1200/JCO.20.00290. Epub 2020 Aug 21. PMID 32822275